CLINICAL TRIAL: NCT01417624
Title: The Assessment of Cardiac Magnetic Resonance Imaging Guided Left Ventricular Lead Placement During the Implantation of Cardiac Resynchronisation Therapy on Clinical Outcomes in Patients With Chronic Heart Failure
Brief Title: Cardiac Magnetic Resonance Imaging Guided Left Ventricular Lead Placement
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Dr Rakesh Sharma, Consulant Cardiologist, Royal Brompton Hospital, Royal Brompton & Harefield NHS Foundation Trust, Sydney Street, London, SW3 6NP, UK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBH2011HS008B
Record Dates: First submitted 2011-08-11; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac Resynchronisation Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group - Standard (Placebo Comparator): This will be a randomised controlled unblinded prospective study recruiting patients in sinus rhythm with LBBB (QRS width ≥ 120ms) and a LV ejection fraction of below 35% who meet the current guidelines for CRT implantation. Patients will be randomised to one of two groups (1:1 randomisation)
  Conventional LV lead placement - the LV lead will be placed according to standard techniques without knowledge of the patient's CMR findings
  Interventions: Other: CMR Guidance in terms of guiding LV lead implantation
- Active CMR guided Arm (Active Comparator): This will be a randomised controlled unblinded prospective study recruiting patients in sinus rhythm with LBBB (QRS width ≥ 120ms) and a LV ejection fraction of below 35% who meet the current guidelines for CRT implantation.Patients will be randomised to one of two groups (1:1 randomisation):
  CMR guided LV lead placement - an expert panel will decide pre-operatively the optimal branch of the coronary sinus for LV lead placement based on the presence of myocardial scar tissue and coronary sinus anatomy. The operator will informed as to the optimal vein to target for delivery of the LV lead. Should this be technically unfeasible (e.g. due to pacing considerations or stability of LV lead position), then the most suitable vein will be used at the time of implantation.
  Interventions: Other: CMR Guidance in terms of guiding LV lead implantation

INTERVENTIONS:
Other: CMR Guidance in terms of guiding LV lead implantation — Following randomisation, the optimal position of the LV lead will be determined either according to current standard criteria (as proposed by the primary operator) or with CMR guidance.
  The CRT device will be implanted using established conventional techniques. The CMR study will be performed pre-implantation only. The distribution of myocardial scar and fibrosis will be derived from this study. A CMR venogram will also be generated and the suggested optimal venous tributaries of the great cardiac vein will be identified from discussion between the principal investigator and senior CMR physician. This information will be used for those in the active arm only.
  Other Names: A cardiac Magnetic resonance Scan using Gadolinium Contrast

SUMMARY:
Heart failure is a common, costly, disabling and potentially lethal condition. Despite well recognised and proven drug therapies, many patients remain breathless on exertion. A special pacemaker (cardiac resynchronisation therapy) may help improve symptoms of breathlessness and survival by restoring coordinated beating of the heart. However, despite careful planning and the knowledge of the most appropriate selection criteria, up to a third of patients do not get the desired beneficial effects after the pacemaker has been implanted.

The implantation of the special pacemaker requires three leads (wires) to be inserted within the heart. Currently this is undertaken under X-ray guidance. Some patients may have scarring of the heart muscle due to previous heart attacks or their underlying condition. The X-ray technique cannot see this and therefore the doctor may implant the lead in such an area of scar tissue. Cardiac magnetic resonance imaging (CMR) can demonstrate these areas of scar. The study aims to investigate whether CMR can better predict where the wires should be placed. The CMR pictures will be taken before the patient has the special pacemaker implanted.

DETAILED DESCRIPTION:
Cardiac Resynchronisation Therapy (CRT) is currently recommended for patients with heart failure who have symptomatic left ventricular (LV) systolic impairment and a prolonged QRS duration.1, 2 Up to a third of patients post CRT implantation do not derive the anticipated clinical benefit. The reasons for this are multifactorial, with patient selection and successful LV lead implantation likely to be key factors.

The mechanism by which CRT exerts its clinical benefits is fundamentally through the correction of mechanical dyssynchrony. However, despite much research in this area the optimal measures of dyssynchrony for the selection of suitable candidates for CRT have not been established. The current guidelines were revised in light of the PROSPECT trial which failed to prove validity and reproducibility in complex echocardiographic variables of dyssynchrony.3 The 12 lead electrocardiogram (ECG) remains the most widely used criterion for the assessment of dyssynchrony in patients being considered for CRT, with patients with a broad QRS complex (>150ms) appearing to benefit the most.4, 5

Although the definition of left bundle branch block (LBBB) is well established, the precise electrophysiological characteristics remain poorly understood. An arbitrary 'cut off' of 120 milliseconds was recommended by the New York Heart Association (NYHA) in 1948 for its definition.6 This has subsequently become enshrined in the literature. The presence of LBBB, a heterogeneous entity, is associated with both electrical and mechanical abnormalities within the left ventricle.7 Septal and lateral wall delay frequently occur in this setting, with delayed activation of the lateral LV wall forming the basis for bi-ventricular pacing. It is well documented within populations with left ventricular impairment that there is prolongation of the QRS complex which is associated with an adverse prognosis.8

The success of CRT is reliant upon achieving an acceptable position of the left ventricular lead during implantation. The LV lead position needs to be anatomically stable to minimise the risk of lead displacement and also to avoid diaphragmatic capture. Furthermore, patients with myocardial scar tissue in the lateral LV segments as detected on CMR are known to have a worse outcome following CRT 9 and pacing such sites may potentially be pro-arrhythmic.10 It is not known whether CMR guided placement of the LV lead in order to avoid sites of myocardial scar and fibrosis can result in an improved clinical outcome in these patients.

A recently published study corroborates that myocardial scar in the region of activation of the LV lead may have a detrimental effect on the delivery of CRT. A consecutive series of 397 patients with ischaemic cardiomyopathy were imaged prior to the implantation of CRT. Using the complex echocardiographic technique of 'speckle tracking', myocardial scar was demonstrated to have an adverse effect on patients' outcomes. It remained an independent predictor of adverse clinical outcome. Notably due to the complexity of the technique, the presence of myocardial scar was validated using CMR.11

CRT response is a contentious subject. It is well recognised within the literature that approximately 30-40% of patients do not appear to improve clinically following CRT implantation.12 However, the inter-study variability of what has been considered as a marker of response has been wide and several different variables have been utilised.13 Several of the studies have also been small, single centre, and non-randomised. There is currently a lack of consensus in what constitutes 'response' vs 'non-response' following CRT, which may be either defined in terms of markers of LV reverse remodelling or changes in the clinical indices of heart failure or a combination of them both. In an effort to rationalise the endpoints of CRT trials, clinical composite scores have been devised inclusive of both imaging based and clinical endpoints. However, the correlation between both LV remodelling and clinical endpoints when compared using correlation coefficients is marginally better than chance. The realisation that clinical improvement post CRT implantation does not necessarily accompany mechanical remodelling has also confused the issue.

Rationale for Study The aim of the present study is to provide pilot data, the results of which should increase our understanding of the mechanisms by which CRT improves clinical outcomes in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent
* Age >18 years old
* Successful CRT implantation (with or without a defibrillator)
* NYHA Class III-IV Heart Failure (or NYHA II with NYHA III/IV symptoms in the preceding 12 months)
* LVEF <35% (Calculated using echocardiography or Cardiac MR) at the time of implantation
* QRS duration > 120ms with Left Bundle Branch Block morphology on ECG
* Sinus Rhythm
* Optimal Tolerated Medical Therapy for Heart Failure

Exclusion Criteria:

* Severe, life threatening non cardiac disease
* Active malignant disease and recent (<5 years) malignant disease
* Prior Heart Transplant
* Recent history of unstable angina, acute coronary syndrome or myocardial infarction within three months of enrollment into the study
* Pregnancy
* Failure to participate in consent process
* Atrial Fibrillation
* Conventional pacemaker in situ
* Heart Failure requiring constant intravenous therapy including diuretics and/or inotropes
* Recent revascularisation procedure i.e. coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) within the last three months
* Contraindications to a CMR study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test Distance | 12 months
  CMR guided LV lead placement during CRT implantation results in improved exercise tolerance at 12 months in patients with heart failure.

SECONDARY OUTCOMES:
Exercise Tolerance (MVO2) | 6, 12 months following CRT Implantation
  Cardiopulmonary Exercise Testing (Peak Oxygen Consumption, MVO2)
Blood Tests - Serum BNP | 1, 6, 12 months following CRT Implantation
  • B Type Natriuretic Peptide (BNP)
Clinical -NYHA Classification | 1, 6, 12 months following CRT
  NYHA Classification
Quality of Life Questionnaires | 1,6,12 months following CRT Implantation
  Euroqol and Minnesota Quality of Life Questionnaires for HF
Echocardiography | 1,6,12 months following CRT Implantation
  LVEF, LVEDD, LVESD, LVESV, LVEDV
Pacing | 1,6,12 months following CRT Implantation
  Level of Bi Ventricular Pacing and atrial and ventricular arrythmia burden
Blood Test -Urate | 1,6,12 months following CRT Implantation
  Serum Urate

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Sharma, MRCP PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, London, United Kingdom

REFERENCES:
- See also: Homepage for Royal Brompton & Harefield NHS Foundation Trust — http://www.rbht.nhs.uk/